CLINICAL TRIAL: NCT04850378
Title: Causes and Prevention of Thromboembolic Disease in Nephrotic Syndrome
Acronym: CAPTAIN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prot-0824-2019
Record Dates: First submitted 2021-04-09; First posted 2021-04-20 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-05

CONDITIONS: Nephrotic Syndrome; Thromboembolic Disease
Keywords: Nephrotic Syndrome; Glomerulonephritis; Hypoalbuminemia; Proteinuria; Thromboembolic Disease; Membranous Nephropathy
MeSH Terms: conditions — Nephrotic Syndrome; Thromboembolism; Glomerulonephritis; Hypoalbuminemia; Proteinuria; Glomerulonephritis, Membranous | interventions — Dalteparin; apixaban

STUDY DESIGN:
Intervention Model Description: An open-label, controlled, non-randomized, interventional clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Coagulation profile in Nephrotic syndrome (No Intervention): Investigation of the biochemical coagulation profile in patients with nephrotic syndrome.
- Nephrotic syndrome (Experimental): Nephrotic patients without diabetes.
  Interventions: Drug: Dalteparin
- Membranous nephropathy and nephrotic syndrome (Experimental): Membranous nephropathy and nephrotic syndrome.
  Interventions: Drug: Apixaban
- Atrial fibrillation (Active Comparator): Atrial fibrillation with no kidney disease.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Dalteparin — Drug: Dalteparin 200 units/kg once a day for 4-7 days.
  Other Names: Fragmin
  Arms: Nephrotic syndrome
Drug: Apixaban — Drug: Apixaban 5 mg twice a day for 4-7 days.
  Other Names: Eliquis
  Arms: Atrial fibrillation; Membranous nephropathy and nephrotic syndrome

SUMMARY:
The study aims to describe the biochemical coagulation profile and investigate the effect of Low molecular weight heparin and Apixaban on this profile in patients with nephrotic syndrome.

DETAILED DESCRIPTION:
The initial part of the study is a prospective cross-sectional study which will describe the biochemical coagulation profile in nephrotic patients. It will include 60 patients with nephrotic syndrome and data from 50 anonymous blood donors matched in age and gender for comparison.

The second part of the study is an open-label, controlled, non-randomized, interventional clinical trial consisting of 3 groups of patients with nephrotic syndrome or atrial fibrillation treated with either Dalteparin or Apixaban. The study participant is expected to be in stable condition after 4 full days of treatment. For administrative reasons, the final biochemical tests are performed on day 4, 5, 6 or 7 described as day 4 in this protocol.

* Group A: Up to 50 patients with nephrotic syndrome treated with injection Dalteparin 200 Units/kg subcutaneous once a day for 4 days
* Group B: 10 patients with nephrotic syndrome and membranous nephropathy treated with Apixaban 5 mg twice daily for 4 days.
* Group C: 10 patients with atrial fibrillation and no kidney disease treated with Apixaban 5 mg twice daily for 4 days.

Patients participating in the initial part of the study will be included in det second part (Group A) if they meet the inclusion criteria. If the patient is diagnosed with membranous nephropathy it is possible to be included in the initial part as well as the second part (Group A and B).

ELIGIBILITY:
Inclusion Criteria: Nephrotic patients - no intervention

* Age 18-79 years
* Estimated Glomerular Filtration Rate (eGFR) > 49 mL/min/1.73 m2
* P-albumin < 30 g/L
* U-Albumin excretion > 2.2 g/day
* Known glomerular disease including membranous nephropathy, which may cause nephrotic syndrome or diagnostically unresolved nephrotic syndrome with a planed kidney biopsy.

Inclusion Criteria: Nephrotic patients treated with Dalteparin

* Age 18-79 years
* eGFR > 49 mL/min/1.73 m2
* P-albumin < 25 g/L
* U-Albumin excretion > 2.2 g/day
* Known glomerular disease including membranous nephropathy, which may cause nephrotic syndrome or diagnostically unresolved nephrotic syndrome with a planed kidney biopsy.

Inclusion Criteria: Nephrotic patients treated with Apixaban

* Age 18-79 years
* eGFR > 49 mL/min/1.73 m2
* P-albumin < 25 g/L
* U-Albumin excretion > 2.2 g/day
* Membranous Nephropathy

Inclusion Criteria: Patients with atrial fibrillation treated with Apixaban

* Age 18-79 years
* eGFR > 49 mL/min/1.73 m2
* P-albumin > 36 g/L
* U-Albumin excretion < 300 mg/day
* Atrial Fibrillation

Exclusion Criteria:

* Contraindication to Apixaban
* Contraindication to Dalteparin
* Known allergy or intolerance to Apixaban
* Known allergy or intolerance to Dalteparin
* Treatment with anticoagulation for other reasons.
* Treatment with cyclooxygenase-1-inhibitors or Adenosine Diphosphate (ADP) receptor inhibitors.
* Known acquired or congenital coagulation defect non related to nephrotic syndrome or thromboembolic disease within 3 months.
* Known diabetes mellitus.
* Lack of compliance, comorbidity or other conditions that, in the patients unfit to participate in the trial.
* Pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Initial Thrombin Generation Assay in nephrotic patients treated with Dalteparin | Predose on Day 1
  Thrombin Generation Assay is used to monitor the anticoagulation therapy
Steady state Thrombin Generation Assay (TGA) in nephrotic patients treated with Dalteparin (Nadir TGA value) | Predose day 4
  Thrombin Generation Assay is used to monitor the anticoagulation therapy
Steady state Thrombin Generation Assay (TGA) in nephrotic patients treated with Dalteparin (4 hours TGA value) | 4 hours postdose on Day 4
  Thrombin Generation Assay is used to monitor the anticoagulation therapy
Initial Thrombin Generation Assay in nephrotic patients treated with Apixaban | Predose on Day 1
  Thrombin Generation Assay is used to monitor the anticoagulation therapy.
Thrombin Generation Assay in nephrotic patients treated with Apixaban over the first 24 hours. | 24 hours
  Thrombin Generation Assay is used to monitor the anticoagulation therapy with blood samples at 2.5, 8, 24 hours.
Steady state Thrombin Generation Assay in nephrotic patients treated with Apixaban. | Predose day 4
  Thrombin Generation Assay is used to monitor the anticoagulation therapy.
Initial Thrombin Generation Assay in patients with atrial fibrillation and no kidney disease treated with Apixaban | Predose on Day 1
  Thrombin Generation Assay is used to monitor the anticoagulation therapy.
Thrombin Generation Assay in patients with atrial fibrillation and no kidney disease treated with Apixaban over the first 24 hours. | 24 hours
  Thrombin Generation Assay is used to monitor the anticoagulation therapy with blood samples at 2.5, 8, 24 hours.
Steady state Thrombin Generation Assay in patients with atrial fibrillation and no kidney disease treated with Apixaban. | Predose day 4
  Thrombin Generation Assay is used to monitor the anticoagulation therapy.
Comparing Thrombin Generation Assay between group B and C. | Predose, 2.5, 8, 24 hours and predose Day 4
  Comparing Thrombin Generation Assay in nephrotic patients treated with Apixaban and patients with atrial fibrillation treated with Apixaban.
Comparing Thrombin Generation Assay between group A and C. | Baseline and predose Day 4
  Comparing Thrombin Generation Assay in nephrotic patients treated with Dalteparin and patients with atrial fibrillation treated with Apixaban.
Comparing Thrombin Generation Assay between group A and B. | Baseline and predose Day 4
  Comparing Thrombin Generation Assay in nephrotic patients treated with Dalteparin and nephrotic patients treated with Apixaban.

SECONDARY OUTCOMES:
Evaluation of bleeding-events durin the study. | Predose until 7 days after last dose of apixaban.
  Number of cases with bleeding-events.
Evaluation of thromboembolic complications during the study. | Predose until 7 days after last dose of apixaban.
  Number of cases with thromboembolic complications
Comparing plasma concentration of Apixaban between group B and C | Day 4
  Comparing plasma-Apixaban in nephrotic patients and patients with atrial fibrillation.
Comparing urine concentration of Apixaban between group B and C | Day 4
  Comparing urine-Apixaban in nephrotic patients and patients with atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kelddal, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelddal S, Grove EL, Duus CL, Nygaard LB, Kristensen T, Mose FH, Gregersen JW, Hvas AM, Birn H. Apixaban Concentrations and Effects on Coagulation in Patients With Nephrotic Syndrome. Kidney Med. 2025 Oct 10;7(12):101136. doi: 10.1016/j.xkme.2025.101136. eCollection 2025 Dec. PMID 41333097
- [Derived] Kelddal S, Grove EL, Duus CL, Nygaard LB, Kristensen T, Mose FH, Gregersen JW, Hvas AM, Birn H. Alterations in Coagulation and Endothelial Function in Nephrotic Syndrome: A Multicenter, Cross-Sectional Analysis. Kidney360. 2025 Nov 1;6(11):1960-1969. doi: 10.34067/KID.0000000865. Epub 2025 Jun 6. PMID 40478760